CLINICAL TRIAL: NCT01048021
Title: Pulmonary Function Changes and Diaphragmatic Paralysis Following Ultrasound Guided Supraclavicular Brachial Plexus Blockade: The Effects of Decreased Local Anesthetic Volume
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Patricia Myktiuk, Dr. Patricia Mykytiuk, University of Manitoba
Other Study IDs: B2008:061
Record Dates: First submitted 2009-11-06; First posted 2010-01-13 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Diaphragmatic Function; Lung Function
Keywords: Measurement of lung mechanics (FEV1, FVC and PEF)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Supraclavicular Block
  Interventions: Procedure: Supraclavicular Block

INTERVENTIONS:
Procedure: Supraclavicular Block — Baseline values of forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and peak expiratory flow rates (PEFR) will be measured in both the sitting and supine position. Ultrasound-guided supraclavicular brachial plexus blocks will be performed in the supine position with a Pajunk 22g block needle and nerve stimulator. The patients will receive local anesthetic injection with 15 mL of 0.75% Bupivicaine. A maximum of 3 cc of 5% Dextrose will be utilized as contrast to confirm needle tip placement and fluid spread prior to injection of the local anesthetic.
  At 60 minutes post-injection, FEV1, FVC, and PEFR measurements will be taken in the sitting and supine position.

SUMMARY:
This clinical trial is being conducted to study lung function and movement of the major muscle involved in breathing (the diaphragm) after a brachial plexus nerve block (nerve "freezing"). The purpose of this study is to find out what effects (good and bad) ultrasound guided nerve freezing has on the movement of the patient's diaphragm and their lung function.

The potential advantage of ultrasound guidance will be a lesser chance of freezing the nerves that innervate the diaphragm and thus having less of an effect on lung function.

DETAILED DESCRIPTION:
The supraclavicular approach to brachial plexus blockade was first described by Kulenkampf in 1911. With classic "blind" techniques, an incidence of pneumothorax has been reported ranging from 0.5-6.0%, limiting its widespread use, despite the belief that the supraclavicular approach is the most consistent, effective technique for anesthetizing the brachial plexus. With the advent of ultrasound guidance and real time visualization this risk has been minimized and a resurgence in utilization of this approach has occurred. Increased block success, diminished performance times, and lower anesthetic volumes have been observed with this technique when compared to nerve stimulator techniques. Despite these advantages, brachial plexus anesthesia above the clavicle is associated with diaphragmatic dysfunction and caution must be demonstrated in patients with respiratory disease. Interscalene brachial plexus blockade has been widely documented to produce a 100% incidence of hemidiaphragmatic paresis and an associated 25% mean reduction in forced vital capacity (FVC) with local anesthetic volumes ranging from 20 - 45mL 8-10, these parameters for supraclavicular brachial plexus blockage are not as well defined. Previous investigations report an incidence of hemidiaphragmatic paresis of 1-75% with supraclavicular brachial plexus blockade. This study will address whether diaphragmatic function and respiratory mechanics can be preserved with lower anesthetic volumes in ultrasound guided supraclavicular brachial plexus blockade.

ELIGIBILITY:
Inclusion Criteria:

* eligible patients undergoing Supraclavicular blockade

Exclusion Criteria:

* < 18 years of age,
* mental illness precluding informed consent,
* infection at the injection site,
* coagulopathy,
* allergy to local anesthetics,
* inability to comprehend English,
* pulmonary disease, and
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pateints at the HSC Pain Management Centre
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 60 minutes
Forced vital capacity (FVC) | 60 minutes
Peak expiratory flow (PEF) | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Mykytiuk, MD, Principal Investigator — Department of Anesthesia, University of Manitoba
Locations (1):
- HSC Pain Management Centre, Winnipeg, Manitoba, Canada